CLINICAL TRIAL: NCT00210080
Title: A Double-Blind, Placebo-Controlled, Parallel Group Study of Uridine 5'-Triphosphate (UTP) Solution for Inhalation as an Adjunct in the Diagnosis of Lung Cancer by Sputum Cytology
Brief Title: A Study to Diagnose Lung Cancer by Sputum Cytology (01-312)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 01-312
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2015-09-04 (Estimated); Status verified 2015-09

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Uridine Triphosphate; Solutions; Inhalation

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: Uridine 5'-Triphosphate (UTP) Solution for Inhalation

SUMMARY:
The primary objective of this study is to determine if more diagnoses of lung cancer are obtained from the cytological evaluation of sputum expectorated following a single inhaled dose of UTP compared to sputum expectorated following a single inhaled dose of placebo in patients suspected of having lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* be suspected of having primary lung cancer based upon chest radiograph(s), CT scan(s), or PET scan(s) and with symptom, risk profile, or history suggestive of malignancy
* have FEV1 greater than or equal to 40% predicted normal for age and height

Exclusion Criteria:

* have obtained a confirmed diagnosis for the current suspicious lung tumor
* have been treated for the current, suspicious tumor except in cases in which the current lesion is the recurrence of the same tumor (same location) for which treatment was administered no less than 180 days prior to screening
* have undergone a bronchoscopic examination or pulmonary fine needle aspiration biopsy within 4 days prior to dosing, or have undergone sputum induction within 3 days prior to dosing

Age Groups: Child, Adult, Older Adult
Enrollment: 700
Dates: Start 2001-04; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Proportion of lung cancers (malignancies) diagnosed by sputum cytology

SECONDARY OUTCOMES:
Proportion of centrally and peripherally located lung cancers diagnosed by sputum cytology;
Proportion of small and large lung cancers diagnosed by sputum cytology;
Proportion of lung cancers of various cell types, stages and resectability diagnosed by sputum cytology;
Wet weight of sputum expectorated;
Macrophage content of sputum

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC